CLINICAL TRIAL: NCT07024316
Title: A Phase I-II, N-of-1, Open-Label, Prospective Study to Evaluate the Efficacy and Safety of ATL-001 in Adult Patients With Congenital Erythropoietic Porphyria (CEP)
Brief Title: A Study to Investigate the Improvement of Photosensitivity in Terms of Skin Lesions Associated With CEP Following Administration of Oral ATL-001 (Ciclopirox Oral Solution) in Participants Aged >18 Years of Age With CEP
Acronym: ATL001-PII-CEP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Atlas Molecular Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATL001-PII-CEP; 1R01FD008540-01 (FDA)
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Congenital Erythropoietic Porphyria (CEP)
MeSH Terms: conditions — Porphyria, Erythropoietic | interventions — Ciclopirox

STUDY DESIGN:
Intervention Model Description: N-of-1, Open-Label, Prospective Study. One group treated with the investigational drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATL-001 (Experimental)
  Interventions: Drug: ATL-001 (Ciclopirox oral solution)

INTERVENTIONS:
Drug: ATL-001 (Ciclopirox oral solution) — Daily administration of oral ATL-001

SUMMARY:
This is a study to investigate the effect of oral ATL-001 (ciclopirox) in CEP (Congenital Erythropoietic Porphyria) patients. During the study, it will be measured the improvement of skin lesions, fatigue and other clinical symptoms as well as blood parameters. Funding source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at the time of signing the informed consent form (ICF)
2. Diagnosis of CEP, based on medical history and/or biochemical porphyrin analysis. Sponsor will review the CEP diagnostic criteria (medical history or biochemical porphyrin analysis) of each potential patient, written Sponsor approval before starting the run-in period will be required
3. a) Female participants must not be pregnant or lactating at screening or admission

3. b) Female participants must be of nonchildbearing potential or agree to use 2 adequate forms of highly effective method(s) of contraception throughout the entire duration of study participation and for at least 4 weeks after the last dose of any study intervention and have negative pregnancy test results at screening (serum) and admission (urine) 4. Male participants with female partners of childbearing potential must be surgically sterile (successful vasectomy at least 4 weeks prior to Day 1) or agree to use adequate forms of highly effective contraception (together with their female partner) for the duration of the study and for at least 4 weeks after the last dose of study intervention; must also agree to refrain from sperm donation during the study and for at least 4 weeks after the last dose of study intervention 5. Negative pregnancy test (females of childbearing potential) at Screening (Month -6), at Baseline (Day 1) and at every visit site until EoS prior to dosing 6. Able to understand the study aims, procedures, and requirements, and provide written informed consent 7. Able to comply with all study procedures 8. Able and committed to complete study patient diaries and questionnaires

Exclusion Criteria:

1. Other than CEP, an inherited or acquired red cell disease associated with anemia
2. Any other photodermatosis such as solar urticaria
3. A history or known allergic reaction to any investigational product excipients or the investigational drug
4. Major surgery within 8 weeks before Screening, incomplete recovery from any previous surgery or planned major surgery during the study
5. History of alcohol dependence or excessive alcohol consumption, as assessed by the Investigator
6. Human immunodeficiency virus (HIV), active Hepatitis B, or C. A positive hepatitis result should be discussed between the Investigator and Sponsor prior to enrolment
7. Score of Personal Health Questionnaire Depression Scale (PHQ-8) ≥10 at screening or any response of "yes" on the Columbia-Suicide Severity Rating Scale (C-SSRS)
8. Uncontrolled medical condition or concomitant medication that would confound the ability to interpret clinical, clinical laboratory, or participant diary data, including a major psychiatric condition that has had an exacerbation or required hospitalization in the last 6 months
9. Administration of afamelanotide and dersimelagon within the last 2 months prior to start of the run-in period
10. Total bilirubin >2× ULN (unless documented Gilbert syndrome) at Screening
11. If female, pregnant or breastfeeding. Final_V2.1 38 of 106 11 Apr 2025
12. Participation in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices within 30 days of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of ATL-001 in patients with CEP in terms of change in lesions associated with photosensitivity. | From Baseline to 12 weeks intervals until the end of study (48 weeks)
  Change between 6-month run-in period and 12-weekly treatment intervals in number and severity of sunlight-induced events measured with the Dermatological Sunlight Questionnaire (DSQ) on a daily basis:
  * Number of lesions
  * Average time to recovery of lesions
  * Number of other symptoms and clinical signs

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinics, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided